CLINICAL TRIAL: NCT05317754
Title: Effectiveness of Four Deconstructive Meditative Practices on Well-being and Self-deconstruction: An Exploratory Randomized Controlled Trial
Brief Title: Effectiveness of Four Deconstructive Meditative Practices on Well-being and Self-deconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI22/110
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Wellness
Keywords: Deconstructive meditation practices; Mindfulness; Randomized controlled trial; Wellbeing; Self-deconstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mindful breathing (Experimental)
  Interventions: Behavioral: Mindful breathing
- Prostrations, according to Tibetan Buddhist tradition (Experimental)
  Interventions: Behavioral: Prostrations, according to Tibetan Buddhist tradition
- The Koan Mu, according to Zen Buddhist tradition (Experimental)
  Interventions: Behavioral: The Koan Mu, according to Zen Buddhist tradition
- The mirror exercise, according to Toltec tradition (Experimental)
  Interventions: Behavioral: The mirror exercise, according to Toltec tradition

INTERVENTIONS:
Behavioral: Mindful breathing — * Formal practice should take 30-60 minutes/day. It can be divided into as many as 4 sessions/day at times of participants' choosing, but the recommended times are after waking up in the morning and before going to bed at night.
  * There is no limit to the number of times informal practice can be performed during the day.
  * Use of a diary is necessary to record the time and duration of all formal and informal practices.
  * The intervention will have a duration of 60 days. During this period, participants are to take part only in the intervention to which they have been randomized and no other. After this period of time and during the follow-up, participants will be able to practise any kind of meditation and at times of their choosing, but this information must always be recorded in their diary.
  Arms: Mindful breathing
Behavioral: Prostrations, according to Tibetan Buddhist tradition — * Formal practice should take 30-60 minutes/day. It can be divided into as many as 4 sessions/day at times of participants' choosing, but the recommended times are after waking up in the morning and before going to bed at night.
  * There is no limit to the number of times informal practice can be performed during the day.
  * Use of a diary is necessary to record the time and duration of all formal and informal practices.
  * The intervention will have a duration of 60 days. During this period, participants are to take part only in the intervention to which they have been randomized and no other. After this period of time and during the follow-up, participants will be able to practise any kind of meditation and at times of their choosing, but this information must always be recorded in their diary.
  Arms: Prostrations, according to Tibetan Buddhist tradition
Behavioral: The Koan Mu, according to Zen Buddhist tradition — * Formal practice should take 30-60 minutes/day. It can be divided into as many as 4 sessions/day at times of participants' choosing, but the recommended times are after waking up in the morning and before going to bed at night.
  * There is no limit to the number of times informal practice can be performed during the day.
  * Use of a diary is necessary to record the time and duration of all formal and informal practices.
  * The intervention will have a duration of 60 days. During this period, participants are to take part only in the intervention to which they have been randomized and no other. After this period of time and during the follow-up, participants will be able to practise any kind of meditation and at times of their choosing, but this information must always be recorded in their diary.
  Arms: The Koan Mu, according to Zen Buddhist tradition
Behavioral: The mirror exercise, according to Toltec tradition — * Formal practice should take 30-60 minutes/day. It can be divided into as many as 4 sessions/day at times of participants' choosing, but the recommended times are after waking up in the morning and before going to bed at night.
  * There is no limit to the number of times informal practice can be performed during the day.
  * Use of a diary is necessary to record the time and duration of all formal and informal practices.
  * The intervention will have a duration of 60 days. During this period, participants are to take part only in the intervention to which they have been randomized and no other. After this period of time and during the follow-up, participants will be able to practise any kind of meditation and at times of their choosing, but this information must always be recorded in their diary.
  Arms: The mirror exercise, according to Toltec tradition

SUMMARY:
The efficacy of interventions based on mindfulness and compassion has been demonstrated in both clinical and general population, and in different social contexts. These interventions include so-called attentional and constructive meditation practices, respectively. However, unlike these, there is a third group, known as deconstructive meditation practices, which has not been scientifically studied. Deconstructive practices aim to undo maladaptive cognitive patterns and generate knowledge about internal models of oneself, others and the world. Although there are theoretical and philosophical studies on the origin of addiction to the self or on the mechanisms of action associated with the deconstruction of the self, there are no randomized controlled trials evaluating these techniques in either a healthy population or clinical samples. This study aims to evaluate the effect of three deconstructive techniques by comparing them to the practice of mindfulness in the general population.

A randomized controlled clinical trial (RCT) will be conducted with about 240 participants allocated (1:1:1:1) to four groups: a) mindful breathing, b) prostrations, according to Tibetan Buddhist tradition; c) the Koan Mu, according to Zen Buddhist tradition; and d) the mirror exercise, according to Toltec tradition. The primary outcome will be the qualities of the non-dual experience and spiritual awakening, measured by the Nondual Embodiment Thematic Inventory, assessed at pre and post-treatment and at 3 and 6-month follow ups. Other outcomes will be mindfulness, happiness, compassion, affectivity and altered state of consciousness. Outcomes at each time point will be compared using mixed-effects linear regression models adjusted for baseline scores, sex and age.

This is the first RCT to apply deconstructive meditation techniques to evaluate their effect on the general population. The positive results of this project may have an important impact on the development of new interventions, not only to improve happiness and well-being in healthy populations but also potentially for the prevention and treatment of psychological and medical disorders, creating a new paradigm in the context of third-generation psychological interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years of age
2. No psychiatric diagnosis (self-reported)
3. More than 1 year's experience of daily meditation practice
4. Having a computer and Internet connection at home
5. Being able to read and understand the Spanish language
6. Willingness to participate in the study and sign the written informed consent form

Exclusion Criteria:

1. Any diagnosis of a disease that may affect the central nervous system (pathological condition affecting the brain, traumatic brain injury, dementia) or other psychiatric diagnoses or acute psychiatric illnesses (severe range of depression, substance dependence or abuse, history of schizophrenia or other psychotic disorders, eating disorders), except for anxiety disorder
2. Any medical, infectious or degenerative disease that may affect mood; presence of delusional ideas; and hallucinations consistent or not with mood and suicide risk
3. Taking any psychiatric medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-11 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Nondual Embodiment Thematic Inventory (NETI) | Baseline
  In the mindful breathing group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Post-treatment 60 days from baseline
  In the mindful breathing group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Three-months follow-up
  In the mindful breathing group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Six-months follow-up
  In the mindful breathing group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Post-treatment 60 days from baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Three-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Six-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Post-treatment 60 days from baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Three-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Six-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Baseline
  In the mirror exercise, according to Toltec tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Post-treatment 60 days from baseline
  In the mirror exercise, according to Toltec tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Three-months follow-up
  In the mirror exercise, according to Toltec tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness
The Nondual Embodiment Thematic Inventory (NETI) | Six-months follow-up
  In the mirror exercise, according to Toltec tradition, group. A total score, ranging from 20 to 100, is calculated by totalling the scores from all the items, with higher scores indicating higher levels of non-dual awareness

SECONDARY OUTCOMES:
Sociodemographic data gender, age, nationality, current city of residence, marital status, education and for information regarding their experience with meditation. | Baseline
  In the mindful breathing group
Sociodemographic data gender, age, nationality, current city of residence, marital status, education and for information regarding their experience with meditation. | Baseline
  In the prostrations, according to Tibetan Buddhist tradition, group
Sociodemographic data gender, age, nationality, current city of residence, marital status, education and for information regarding their experience with meditation. | Baseline
  In the Koan Mu, according to Zen Buddhist tradition, group
Sociodemographic data gender, age, nationality, current city of residence, marital status, education and for information regarding their experience with meditation. | Baseline
  In the mirror exercise, according to Toltec tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Baseline
  In the mindful breathing group
The Nondual Awareness Dimensional Assessment (NADA) | Post-treatment 60 days from baseline
  In the mindful breathing group
The Nondual Awareness Dimensional Assessment (NADA) | Three-months follow-up
  In the mindful breathing group
The Nondual Awareness Dimensional Assessment (NADA) | Six-months follow-up
  In the mindful breathing group
The Nondual Awareness Dimensional Assessment (NADA) | Baseline
  In the prostrations, according to Tibetan Buddhist tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Post-treatment 60 days from baseline
  In the prostrations, according to Tibetan Buddhist tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Three-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Six-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Baseline
  In the Koan Mu, according to Zen Buddhist tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Post-treatment 60 days from baseline
  In the Koan Mu, according to Zen Buddhist tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Three-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Six-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Baseline
  In the mirror exercise, according to Toltec tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Post-treatment 60 days from baseline
  In the mirror exercise, according to Toltec tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Three-months follow-up
  In the mirror exercise, according to Toltec tradition, group
The Nondual Awareness Dimensional Assessment (NADA) | Six-months follow-up
  In the mirror exercise, according to Toltec tradition, group
The Five Facet Mindfulness Questionnaire (FFMQ) | Baseline
  In the mindful breathing group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Post-treatment 60 days from baseline
  In the mindful breathing group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Three-months follow-up
  In the mindful breathing group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Six-months follow-up
  In the mindful breathing group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Post-treatment 60 days from baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Three-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Six-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Post-treatment 60 days from baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Three-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Six-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Baseline
  In the mirror exercise, according to Toltec tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Post-treatment 60 days from baseline
  In the mirror exercise, according to Toltec tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Three-months follow-up
  In the mirror exercise, according to Toltec tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
The Five Facet Mindfulness Questionnaire (FFMQ) | Six-months follow-up
  In the mirror exercise, according to Toltec tradition, group. A total score, ranging from 39 to 195, is calculated by totalling the scores from all the items, and higher total values indicate better full mindfulness
Sussex-Oxford Compassion Scales (SOCS) | Baseline
  In the mindful breathing group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Post-treatment 60 days from baseline
  In the mindful breathing group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Three-months follow-up
  In the mindful breathing group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Six-months follow-up
  In the mindful breathing group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Post-treatment 60 days from baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Three-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Six-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Post-treatment 60 days from baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Three-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Six-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Baseline
  In the mirror exercise, according to Toltec tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Post-treatment 60 days from baseline
  In the mirror exercise, according to Toltec tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Three-months follow-up
  In the mirror exercise, according to Toltec tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
Sussex-Oxford Compassion Scales (SOCS) | Six-months follow-up
  In the mirror exercise, according to Toltec tradition, group. This scale is composed by two 20-item self-report scales measuring compassion. A total score, ranging from 20 to 100, is calculated for each scale, and higher total values indicate higher levels of compassion
The Pemberton Happiness Index (PHI) | Baseline
  In the mindful breathing group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Post-treatment 60 days from baseline
  In the mindful breathing group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Three-months follow-up
  In the mindful breathing group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Six-months follow-up
  In the mindful breathing group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Post-treatment 60 days from baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Three-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Six-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Post-treatment 60 days from baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Three-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Six-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Baseline
  In the mirror exercise, according to Toltec tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Post-treatment 60 days from baseline
  In the mirror exercise, according to Toltec tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Three-months follow-up
  In the mirror exercise, according to Toltec tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
The Pemberton Happiness Index (PHI) | Six-months follow-up
  In the mirror exercise, according to Toltec tradition, group. To calculate the overall PHI index, which included remembered and experienced well-being, individuals' scores of the 11 items related to remembered well-being plus the sum of scores on the experienced well-being were summed; the total sum is then divided by 12, so the resulting PHI total mean score also ranges from 0 to 10. Higher total values indicate higher levels of well-being
Positive and Negative Affect Schedule (PANAS) | Baseline
  In the mindful breathing group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Post-treatment 60 days from baseline
  In the mindful breathing group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Three-months follow-up
  In the mindful breathing group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Six-months follow-up
  In the mindful breathing group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Post-treatment 60 days from baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Three-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Six-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Post-treatment 60 days from baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Three-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Six-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Baseline
  In the mirror exercise, according to Toltec tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Post-treatment 60 days from baseline
  In the mirror exercise, according to Toltec tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Three-months follow-up
  In the mirror exercise, according to Toltec tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Positive and Negative Affect Schedule (PANAS) | Six-months follow-up
  In the mirror exercise, according to Toltec tradition, group. This questionnaire comprises 20 items and two independent dimensions: positive affect and negative effect. Each scale has 10 items, and the score range for each is from 10 to 50. Higher total values indicate higher level of positive affect and negative effect respectively.
Altered state of consciousness rating scale (OAV) | Baseline
  In the mindful breathing group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Post-treatment 60 days from baseline
  In the mindful breathing group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Three-months follow-up
  In the mindful breathing group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Six-months follow-up
  In the mindful breathing group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Post-treatment 60 days from baseline
  In the prostrations, according to Tibetan Buddhist tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Three-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Six-months follow-up
  In the prostrations, according to Tibetan Buddhist tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Post-treatment 60 days from baseline
  In the Koan Mu, according to Zen Buddhist tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Three-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Six-months follow-up
  In the Koan Mu, according to Zen Buddhist tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Baseline
  In the mirror exercise, according to Toltec tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Post-treatment 60 days from baseline
  In the mirror exercise, according to Toltec tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Three-months follow-up
  In the mirror exercise, according to Toltec tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.
Altered state of consciousness rating scale (OAV) | Six-months follow-up
  In the mirror exercise, according to Toltec tradition, group. The items are scored by measuring the millimeters from the low end of the scale to the subject's mark (integers from 0-100). Higher values indicate higher perception of an altered state of consciousness.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry. Miguel Servet University Hospital, Zaragoza, Zaragoza, Spain

REFERENCES:
- [Derived] Garcia-Campayo J, Hijar-Aguinaga R, Lopez-Del-Hoyo Y, Magallon-Botaya R, Fernandez-Martinez S, Barcelo-Soler A, Soler-Ribaudi J, Montero-Marin J. Effectiveness of four deconstructive meditative practices on well-being and self-deconstruction: study protocol for an exploratory randomized controlled trial. Trials. 2023 Feb 20;24(1):125. doi: 10.1186/s13063-023-07151-0. PMID 36805694